CLINICAL TRIAL: NCT03495479
Title: Phase IIA, Single-Center, Single-Arm Clinical Study of OMN54 (Aneustat) in Men Diagnosed With Prostate Cancer Being Followed by Active Surveillance
Brief Title: Aneustat Treatment of Localized Prostate Cancer Under Active Surveillance
Acronym: CAMPAS
Status: Withdrawn | Type: Observational
Why Stopped: No funding
Sponsor: Omnitura Therapeutics, Inc. (Industry)
Collaborators: Vancouver Prostate Centre (Other)
Responsible Party: Sponsor
Other Study IDs: OMN54-PC-02
Record Dates: First submitted 2016-06-14; First posted 2018-04-12 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; PC; Active Surveillance; Chemonaiive; OMN54; Aneustat (TM); PSA; BPH
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- OMN54 -Treated: Six-month, daily oral dosing in softgel capsules throughout the first 6 months of treat.
  Interventions: Drug: OMN54

INTERVENTIONS:
Drug: OMN54 — Twice daily, self administered, oral dosing of OMN54. A daily diary log will be prepared by each participant and reviewed by the Investigator.
  Other Names: Aneustat(TM)

SUMMARY:
Assessment of the effects of OMN54 (Aneustat) in a population of men with indolent prostate cancer who are otherwise healthy and free of significant co-morbidities and have chosen active surveillance for disease management. The investigators will assess how OMN54 affects PSA, overall tumor burden in addition to any changes in urinary flow. Other biomarkers will be tested to follow disease evolution.

ELIGIBILITY:
Inclusion Criteria:

- Localized prostate cancer suitable for active surveillance

1. Histologically confirmed adenocarcinoma of the prostate, with Gleason Score 6 or less prostate cancer. No limit in the percentage of cancer in each core or percentage of positive cores.
2. Male, 18 years or older
3. Able to swallow the soft gelatin capsule form of the drug which is ~6mm long.
4. Clinically localized prostate cancer: T1-2, NX or N0, MX or M0.
5. No previous treatment for prostate cancer (including hormonal therapy, radiation therapy, surgery, or chemotherapy).
6. ECOG Performance Status 0 or 1.
7. Patient has elected Active Surveillance as preferred management plan for prostate cancer.
8. Written informed consent obtained prior to any patient participation.
9. Participant is accessible and compliant for follow-up.
10. Prostate biopsy requirements:

    1. If diagnosis was within one year of baseline visit, participant must have at least one biopsy with at least 10 cores.
    2. If diagnosis was more than 1 year prior to baseline visit, participant must have a minimum of 2 biopsies, one of which must be within 2 years prior to baseline visit.
11. Voiding requirements: IPSS score of at least 15 and Qmax < 15 cc/s.
12. Adequate hematopoietic function as demonstrated by:

    * hemoglobin of ≥ 9.0 g/dL without need for sustained blood transfusions
    * Platelet count ≥100,000 platelet/mm3 (100 x 109/L)
    * White Blood Cell (WBC) count ≥ 2.0 x109/L and Absolute Neutrophil Count (ANC) ≥1.5 x109/L
13. Adequate hepatobiliary function as demonstrated by:

    * Total bilirubin level within normal limits
    * Alanine aminotransferase (ALT) levels within normal limits
    * Adequate renal function as demonstrated by creatinine level within normal limits or creatinine clearance within normal limits
    * Coagulation profile (PT, PTT, INR and TCT) within normal limits
14. If of reproductive capacity, willing to use an effective double barrier method of birth control (i.e., latex condom, partner use of diaphragm, cervical cap, etc) during the study and for 30 days after the last administration of OMN54

Exclusion Criteria:

1. Unwillingness or inability to undergo serial prostate biopsy or MRI.
2. History of other malignancies, except: adequately treated non-melanoma skin cancer or adequately treated superficial bladder cancer (Ta) or other solid tumors curatively treated with no evidence of disease for > 5 years.
3. Previous surgical intervention for BPH
4. Active uncontrolled infection, including known history of HIV, hepatitis B or C
5. Concurrent uncontrolled hypertension
6. Congestive Heart Failure
7. Hepatic disease (cirrhosis, hepatitis, hepatocellular carcinoma or liver failure of unknown etiology)
8. Renal disease (glomerulonephritis, nephropathy, polycystic kidney disease)
9. Patients requiring new treatment of BPH (either medical or surgical) are not eligible.
10. Refractory nausea and vomiting, chronic gastrointestinal diseases (e.g., inflammatory bowel disease), or significant bowel resection that would preclude adequate absorption.
11. Known hypersensitivity to any of the three botanical constituents of Aneustat™ (OMN54); soy; any of the plants belonging to the Ganodermataceae family, e.g., reishi mushroom (Ganoderma lucidum, lingzhi); any plants belonging to Labiatae or Lamiaceae families, e.g., culinary herbs including basil, mint, rosemary, sage, savory, marjoram, oregano, thyme, lavender, and perilla; or Aneustat™ (OMN54) excipients.
12. Concurrent administration, or exposure within 30 days, of:

    * Investigational drugs and devices
    * Chemotherapy
    * Radiation therapy
    * Immunotherapy

Ages: 18 Years to 72 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men diagnosed with early stage prostate cancer that elect to pursue active surveillance for disease management and agree to take the study drug.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Prostate Specific Antigen | 12 months
  Quarterly assessment of serum Prostate Specific Antigen (PSA)
Changes in Tumor Size | 12 months
  Changes in tumor size based on semi-annual MRI
Changes in Urinary Flow | 12 months
  Quartelry assessment of patient urinary flow based on patient IPSS Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Alan So, MD, Principal Investigator — Prostate Centre at Vancouver General Hospital

IPD SHARING:
Plan to Share IPD: Undecided
This is undecided and will be decided in consultation with the PI.